CLINICAL TRIAL: NCT01095016
Title: An Open-label, Randomized, Cross-over, Active-controlled Study to Evaluate the Efficacy and Safety of Meptin® Swinghaler and Berotec N® Metered Aerosol in Mild to Moderate Stable Asthma Patients
Brief Title: A Study to Evaluate the Efficacy and Safety of Meptin® Swinghaler and Berotec N® Metered Aerosol in Mild to Moderate Stable Asthma Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taiwan Otsuka Pharm. Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 002-TWB-0901
Record Dates: First submitted 2010-03-15; First posted 2010-03-29 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Fenoterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Meptin swinghaler (Experimental)
  Interventions: Drug: Meptin swinghaler
- Berotec (Active Comparator)
  Interventions: Drug: Berotec

INTERVENTIONS:
Drug: Meptin swinghaler — * Dose: 10ug/puff, 2 puffs daily
  * Frequency: QD (total 20ug/day)
  * Treatment duration: 2 days
  Arms: Meptin swinghaler
Drug: Berotec — * Dose: 100ug/puff, 2 puffs daily
  * Frequency: QD (total 200ug/day)
  * Treatment duration: 2 days
  Arms: Berotec

SUMMARY:
This is an open-label, randomized, cross-over, active-controlled study to evaluate the efficacy and safety effects using Meptin® Swinghaler and Berotec N® Metered Aerosol in stable asthma patients

ELIGIBILITY:
Inclusion Criteria:

* Male or females outpatients aged ≥18 years old with uncontrolled or partly controlled asthma; Stability was assessed during the past 14 days the patients remained in the same severity class by 2006 GINA guideline (uncontrolled, partly controlled) and had no acute exacerbations by investigator judgment;
* Pulmonary function test: Improvement ≥12% reversibility in FEV1 or FVC following administration of an inhaled β2-agonist before the study or ; Positive result of Brocho-provocation test;

Exclusion Criteria:

* Hypersensitivity to β2-agonist or lactose;
* Hospitalization due to asthma during the previous 3 months;
* Respiratory tract infection requiring treatment with antibiotics in the previous 4 weeks;
* Oral or systemic corticosteroids in the previous 4 weeks;
* Inadequately controlled hyperthyroidism;
* Subjects with any clinically significant disorder of the cardiovascular, neurologic, hematologic, gastrointestinal, cerebrovascular, or immunologic system or respiratory disease other than asthma(e.g. COPD), or any other disorder which may interfere wth the study evaluations or affect subject safety;
* Patients receive an investigational drug within 30 days prior to admission to the study;
* Patients with significant alcohol, drug or medication abuse as judged by the investigator;
* Females who are pregnant or breast-feeding; (exception: Females of child-bearing age might be included, if in the opinion of the investigator, they are using adequate contraceptive precautions);
* Subjects who are heavy smoker (more than 10 packs year) or who are smoking within previous 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The change of Forced Expiratory Volume in 1 second (FEV1) value | 12 months

SECONDARY OUTCOMES:
The change of Peak Expiratory Flow Rate (PEFR) | 12 months
The change of Forced Vital Capacity (FVC) | 12 months
Device acceptance | 12 months
  5-point score of evaluation form to test preference on Meptin swinghaler/ Berotec device by investigator or patient

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hsiu Chung, MD, Principal Investigator — Chang Cung Memorial Hospital
Locations (1):
- Chang Cung Memorial Hospital, Taipei, Taiwan